CLINICAL TRIAL: NCT00958217
Title: Intervention for Veterans With Depression, Substance Disorder, and Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHBA-016-09S
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Depressive Symptoms; Substance-related Disorders; Posttraumatic Stress Disorders
Keywords: Depressive symptoms; Substance-related disorders; Posttraumatic stress disorders; Psychotherapy
MeSH Terms: conditions — Depression; Substance-Related Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive Processing Therapy-Modified (Experimental): 12 individually delivered sessions of Cognitive Processing Therapy-Modified (CPT-M) provided once weekly following initial group delivery of 12 sessions of Integrated Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Processing Therapy-Modified (CPT-M)
- Integrated Cognitive Behavioral Therapy (Active Comparator): 12 individually delivered sessions of Integrated Cognitive Behavioral Therapy (ICBT) once weekly following initial group delivery of 12 sessions of ICBT
  Interventions: Behavioral: Integrated Cognitive Behavioral Therapy (ICBT)
- Integrated Cognitive Behavioral Group Therapy (No Intervention): All participants were enrolled in an initial group-delivered Integrated Cognitive Therapy Group, consisting of 12 sessions over approximately 12 weeks prior to randomization to one of the study individually delivered interventions (CPT-M or ICBT). Individuals who were no longer participating in the study at the end of group sessions were not randomized.

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy-Modified (CPT-M) — Psychotherapy that focuses on thoughts associated with traumatic experiences with the goal of developing skills to reduce trauma-related symptoms. We have modified this therapy to include substance relapse prevention skills, reduce depression and substance relapse. CPT-M was delivered in individual 1-hour sessions once weekly.
  Arms: Cognitive Processing Therapy-Modified
Behavioral: Integrated Cognitive Behavioral Therapy (ICBT) — Psychotherapy that focuses on thoughts and behaviors associated with depression with the goal of developing skills to reduce depression symptoms. We have integrated substance relapse prevention skills. ICBT was delivered in individual 1-hour sessions once weekly.
  Arms: Integrated Cognitive Behavioral Therapy

SUMMARY:
This study will compare two different types of psychotherapy for Veterans with depression, addiction, and a past traumatic experience. Everyone in the study will receive 12 weeks of group cognitive behavioral therapy focused on depression and addiction, followed by 12 weeks of individual psychotherapy sessions. For the second 12 weeks, half of the people will receive a review of the initial therapy, and half will receive a cognitive behavioral therapy focused on trauma. Everyone will complete research interviews every 3 months for a total of 18 months.

DETAILED DESCRIPTION:
The goal of this study is to evaluate whether a second disorder-specific intervention improves longer term (up to 18 months) treatment outcomes for male and female Veterans with co-occurring depression and alcohol/substance disorders and trauma history (with or without PTSD diagnosis). This 4 years randomized two-group design uses repeated assessments at baseline and every 3 months for a total of 12 months. The investigators are providing their recently developed integrated intervention for comorbid depression and substance disorders for the initial 12 weeks in group format (Integrated Cognitive Behavioral Therapy; Phase I). After the 12 week group intervention, participants will be randomized to receive either a review of the initial intervention in individual sessions, or a trauma-specific intervention, Cognitive Processing Therapy, with integrated addiction treatment components. Length, duration, and setting of both interventions will be the same, and all participants will meet with the program psychiatrist for medication appointments. No medications are under study and no placebo is used; medications will be prescribed using standard VA protocol. Research assessments will document diagnosis, recent substance use, depression and PTSD symptoms, medication adherence, and life stress.

ELIGIBILITY:
Inclusion Criteria:

* Veterans 18 years of age and older living in the San Diego, California area
* Who are able to attend in-person therapy sessions
* Have depression, alcohol or substance addiction, and a past traumatic experience

Exclusion Criteria:

* Non-veterans
* Individuals with schizophrenia or severe memory impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Tate, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego/University of California, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Siegel EY, Haller M, Cui R, Trim RS, Tate SR, Norman SB. Examining changes in negative mood regulation expectancies, posttraumatic stress disorder, depression, and substance use following integrated cognitive-behavioral therapy. Subst Abus. 2017 Oct-Dec;38(4):468-472. doi: 10.1080/08897077.2017.1342736. Epub 2017 Jun 20. PMID 28632462
- [Derived] Cui R, Haller M, Skidmore JR, Goldsteinholm K, Norman S, Tate SR. Treatment Attendance Among Veterans With Depression, Substance Use Disorder, and Trauma. J Dual Diagn. 2016;12(1):15-26. doi: 10.1080/15504263.2016.1146384. PMID 26828770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans referred to a VA dual diagnosis outpatient clinic who were diagnosed with depressive disorder, substance use disorder, and had a history of trauma (with and without a posttraumatic stress disorder diagnosis) were recruited from December 2009 through October 2012.
Pre-assignment Details: All participants engaged in 12 weeks of group Integrated Cognitive Behavioral Therapy and were then randomized to the individual study interventions. 31 participants were not randomized (3 died, 6 moved, 6 withdrew, 4 lost, 4 not stable, 4 did not meet study criteria, 4 sober living facility did not allow).
Groups:
- Arm 1: Cognitive Processing Therapy- Modified: Individuals with depression and substance disorders and trauma history (with and without PTSD diagnosis) are randomized to receive one of two psychotherapy interventions.
  CPT-M: Cognitive Processing Therapy-Modified: Psychotherapy that focuses on thoughts associated with traumatic experiences with the goal of developing skills to reduce trauma-related symptoms. We have modified this therapy to include substance relapse prevention skills.
- Arm 2: Integrated Cognitive Behavioral Therapy: Individuals with depression and substance disorders and trauma history (with and without a PTSD diagnosis) are randomized to receive one of two psychotherapy interventions.
  ICBT: Integrated Cognitive Behavioral Therapy: Psychotherapy that focuses on thoughts and behaviors that are associated with depression and substance relapse with the goal of developing skills to reduce depression and substance relapse
Period: Overall Study
Arm/Group | Arm 1: Cognitive Processing Therapy- Modified | Arm 2: Integrated Cognitive Behavioral Therapy
Started | 61 | 62
End of Treatment | 56 (Participants had a maximum of 16 weeks to complete 12 individual psychotherapy sessions) | 57 (Participants had a maximum of 16 weeks to complete 12 individual psychotherapy sessions)
Completed | 37 (Participants were assessed quarterly for one year following end of treatment) | 37 (Participants were assessed quarterly for one year following end of treatment)
Not Completed | 24 | 25
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 17 | 19
Not completed — Moved out of area | 1 | 1
Not completed — Inpatient hospitalization | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: CPT-M: Individuals with depression and substance disorders and trauma history (with and without PTSD diagnosis) were recruited.
  CPT-M: Cognitive Processing Therapy-Modified: Psychotherapy that focuses on thoughts associated with traumatic experiences with the goal of developing skills to reduce trauma-related symptoms. We have modified this therapy to include substance relapse prevention skills.
- Arm 2: ICBT: Individuals with depression and substance disorders and trauma history (with and without a PTSD diagnosis) were recruited.
  ICBT: Integrated Cognitive Behavioral Therapy: Psychotherapy that focuses on thoughts and behaviors that are associated with depression and substance relapse with the goal of developing skills to reduce depression and substance relapse
- Total: Total of all reporting groups
Arm/Group | Arm 1: CPT-M | Arm 2: ICBT | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (12.1) | 47.3 (11.9) | 47.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 55 | 54 | 109
PTSD Current diagnosis [Number; unit: participants]
  with PTSD diagnosis | 51 | 50 | 101
  without PTSD diagnosis | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Depression Symptoms Were Assessed With the Hamilton Depression Rating Scale.
Description: Depression symptoms were assessed using a structured clinical interview assessment consisting of 21 items. Depression symptoms experienced in the past week are rated on a 0 (none) to 4 (most severe) scale. The total score is summed from the item scores and range from 0 (none) to 84 (most severe). We tested whether treatment group interacted with time in order to examine whether trajectories of symptom scores differed across treatment conditions. Linear mixed effects models were used to ascertain trajectories of total scores from randomization through end of study (6 timepoints across approximately 15 months). This analytic approach was advantageous in that it provided examination of change in depression across all quarterly assessments. Models were estimated with maximum likelihood methods. Total score at the time of randomization is reported in Data Table and coefficient estimates for trajectories are reported in Statistical Analysis.
Time Frame: Assessed quarterly; trajectories analyzed total scores from randomization through end of study (6 timepoints covering approximately 15 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Cognitive Processing Therapy- Modified | Arm 2: Integrated Cognitive Behavioral Therapy
Number analyzed (Participants) | 61 | 62
units on a scale | 31.92 (12.37) | 28.85 (12.25)
Statistical Analysis 1: Comparison: Arm 1: Cognitive Processing Therapy- Modified vs Arm 2: Integrated Cognitive Behavioral Therapy; Data analyses included comparison of mean scores and linear mixed effects models used to ascertain trajectories for depression symptoms; Test type: Superiority or Other; p < .05, Linear Mixed Effects Models — P-values based on likelihood ratio tests for the significance of the first and second order trajectory parameters. Primary tests compared curvilinear trajectories of the two treatment groups; 2nd order effects of time (2 slope = 33 — We gauged sampling error with 95% confidence bands

2. Primary Outcome: Posttraumatic Stress Disorder (PTSD) Symptoms
Description: The Posttraumatic Stress Disorder Checklist - Civilian version (PCL-C) is a 17 item self-report checklist of PTSD symptoms experienced in the past month rated on a 1 (not at all) to 5 (extremely) scale; total score is summed from the item scores and range from 17 (none) to 85 (most severe). . Civilian version was selected as it allows for a variety of trauma types. Scores above 50 are considered clinical levels. We tested whether treatment group interacted with time to examine whether trajectories of symptom scores differed across treatment conditions. Linear mixed effects models were used to ascertain trajectories of total scores. This analytic approach was advantageous in that it provided examination of change in PTSD across all quarterly assessments. Models were estimated with maximum likelihood methods. Total score at the time of randomization is reported in Data Table and coefficient estimates for trajectories are reported in Statistical Analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Cognitive Processing Therapy- Modified | Arm 2: Integrated Cognitive Behavioral Therapy
Number analyzed (Participants) | 61 | 62
units on a scale | 58.4 (12.4) | 55.5 (14.2)
Statistical Analysis 1: Comparison: Arm 1: Cognitive Processing Therapy- Modified vs Arm 2: Integrated Cognitive Behavioral Therapy; Test type: Superiority or Other; p < .05, Linear Mixed Effects Models; Second order effect of time (2 slopes) = 57.0 — We gauged sampling error with 95% confidence bands

3. Primary Outcome: Timeline Followback
Description: The Timeline Followback is a calendar-assisted structured interview that assesses the frequency of alcohol and drug use on a daily basis and the quantity of alcohol use. Summary proportion of days abstinent were calculated at each time point. Trajectory analyses examine two substance use outcomes: probability of any alcohol or drug use on a given day and probability of heavy drinking (5 or more drinks consumed in a day) on a given day. Trajectories of substance use (any alcohol or drug use on a particular day) and heavy drinking (>5 drinks on a particular day) were modeled as dichotomous outcomes, using logit links to predict the probability of substance use or heavy drinking on a particular day. Data Table reports starting proportion of days abstinent at time of randomization.
Time Frame: Assessed quarterly; trajectories analyzed from randomization through end of study (covering approximately 15 months)
Measure: Mean (Standard Deviation); unit: proportion of days abstinent
Arm/Group | Arm 1: Cognitive Processing Therapy- Modified | Arm 2: Integrated Cognitive Behavioral Therapy
Number analyzed (Participants) | 61 | 62
proportion of days abstinent | .84 (.26) | .81 (.30)
Statistical Analysis 1: Comparison: Arm 1: Cognitive Processing Therapy- Modified vs Arm 2: Integrated Cognitive Behavioral Therapy; Analysis of substance use was conducted using trajectories modeled as a dichotomous outcome using logit links to predict the probability of substance use (any alcohol or drug use) on a particular day; Test type: Superiority or Other; p < .05, Linear Mixed Effects Model; A logit link was used in this model; Second order effect of time (2 slopes) = .43 — We gauged sampling error with 95% confidence bands
Statistical Analysis 2: Comparison: Arm 1: Cognitive Processing Therapy- Modified vs Arm 2: Integrated Cognitive Behavioral Therapy; Second statistical analysis evaluates trajectories of heavy drinking (<5 drinks on a given day) Analysis of heavy drinking was conducted using trajectories modeled as a dichotomous outcome using logit links to predict the probability of heavy drinking (5 or more drinks) on a particular day; Test type: Superiority or Other; p < .05, Linear Mixed Effects Model; A logit link was used in this model; Second order effect of time (2 slopes) = .26 — We gauged sampling error with 95% confidence bands

ADVERSE EVENTS:
Time Frame: 4 years
Description: Number at Risk for Serious Adverse Events in the ICBT Prior to Randomization Arm is 23, excluding 4 participants who were lost and 4 participants who did not meet study criteria; we have no data and Adverse Events were not collected for these 8. For Other Adverse Events, we excluded 3 participants who died and not at risk for events.
Groups:
- ICBT Prior to Randomization: All participants attended 12 weeks of group Integrated Cognitive Behavioral Therapy prior to randomization to provide for a period of stabilization and to develop relapse prevention and mood management skills.
  This portion will report on only those participants who were not randomized to individual CPT-M or ICBT.
Arm/Group | Arm 1: Cognitive Processing Therapy- Modified | Arm 2: Integrated Cognitive Behavioral Therapy | ICBT Prior to Randomization
Serious Adverse Events (participants affected / at risk) | 15/61 | 19/62 | 10/23
Other Adverse Events (participants affected / at risk) | 25/61 | 55/62 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Cognitive Processing Therapy- Modified (N=61) | Arm 2: Integrated Cognitive Behavioral Therapy (N=62) | ICBT Prior to Randomization (N=23)
Inpatient psychiatric admission for suicidal ideation/behaviors (Psychiatric disorders) | 6 | 10 | 3
Inpatient admission for alcohol/drug treatment (Psychiatric disorders) | 4 | 1 | 1
Death - unknown cause (General disorders) | 1 | 0 | 3
Death - liver disease (Hepatobiliary disorders) | 1 | 0 | 0
Death - hit by motor vehicle (Injury, poisoning and procedural complications) | 0 | 1 | 0
Suicidal behavior under the influence (Psychiatric disorders) | 0 | 1 | 0
Medical inpatient admission - alcohol related (Gastrointestinal disorders) | 1 | 2 | 1
Medical inpatient admission - infection (Infections and infestations) | 1 | 3 | 0
Medical inpatient admission - surgery (Gastrointestinal disorders) | 0 | 0 | 1
Medical inpatient admission - assault injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Disappearance (Psychiatric disorders) | 0 | 1 | 0 — Left sober living facility and left all belongings without notice and no information
Emergency Dept visit - intoxication (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Cognitive Processing Therapy- Modified (N=61) | Arm 2: Integrated Cognitive Behavioral Therapy (N=62) | ICBT Prior to Randomization (N=20)
Arrest/jail/legal (Psychiatric disorders) | 6 (6) | 10 (10) | 1 (1) — Arrests, brief incarceration, or court appearances related to alcohol/drug use
Outpatient surgery (General disorders) | 1 (1) | 10 (10) | 0 (0) — Outpatient surgeries for variety of medical issues
Urgent Care, Medical (General disorders) | 15 (15) | 32 (32) | 0 (0) — Emergency Department or Urgent Care treatment for variety of medical issues
Urgent Care, Psychiatric (Psychiatric disorders) | 3 (3) | 3 (3) | 0 (0) — Emergency Department or Urgent Care treatment for psychiatric and substance-related issues

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No